CLINICAL TRIAL: NCT03751579
Title: Validation of the Respiratory Quotient Measurement Measured Indirectly in Coelioscopic Surgery
Brief Title: Indirect Measurement of Respiratory Quotient in Coelioscopic Surgery
Status: Withdrawn | Type: Observational
Why Stopped: no participant enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0046
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Quotient Measurement
Keywords: coelioscopic; surgery complications; respiratory quotient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: coelioscopic surgery — observational study based on the computation of respiratory quotient in patient cohort treated by routine coelioscopic surgery

SUMMARY:
The measurement of VO2 and VCO2 makes it possible to calculate the respiratory quotient (RQ) (VCO2 / VO2) which is a reflection of human energy metabolism and therefore of anaerobiosis. A study has been conducted in our department to demonstrate the ability of the indirectly measured RQ from the inspired and exhaled breath analysis of the anesthetic respirator to predict the onset of anaerobic metabolism and postoperative complications in the operating room.

But, because of artificially increase of carbon dioxide due to insufflation, coelioscopic surgery was an exclusion criteria of our pilot study.

However, no study has examined the impact of coelioscopy on the indirect measurement of RQ

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Adults admitted to the operating room for coelioscopic surgery

Exclusion Criteria:

* Cardiac and thoracic surgery
* Preoperative oxygen therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Age>18 years old
  * Adults admitted to the operating room for coelioscopic surgery
  Exclusion Criteria:
  * Cardiac and thoracic surgery
  * Preoperative oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Indirect respiratory quotient by measurement of VO2 and VCO2 | during coelioscopic surgery
  The measurement of VO2 and VCO2 makes it possible to calculate the respiratory quotient (RQ) (VCO2 / VO2)

SECONDARY OUTCOMES:
occurence of at least one post-operative complication | through study completion, an average of 6 months
  the aim is to predict the occurence of at least one complication with the use of indirect respiratory quotient

REFERENCES:
- [Derived] Bar S, Santarelli D, de Broca B, Abou Arab O, Leviel F, Miclo M, Dupont H, Guinot PG, Lorne E. Predictive value of the respiratory exchange ratio for the occurrence of postoperative complications in laparoscopic surgery: a prospective and observational study. J Clin Monit Comput. 2021 Aug;35(4):849-858. doi: 10.1007/s10877-020-00544-5. Epub 2020 Jun 12. PMID 32533528